CLINICAL TRIAL: NCT02790112
Title: Influence of Early Adiposity Rebound, Genetic Polymorphisms and GnRHa Treatment on Long-term Outcome of Girls With Idiopathic Central Precocious Puberty.
Brief Title: Long-term Outcome of GnRH Analogues Treatment of Children With Idiopathic Central Precocious Puberty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Belgian Study Group for Pediatric Endocrinology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2015/14OCT/549; RESEARCH GRANT (Other Grant/Funding Number: BELGIAN STUDY GROUP FOR PEDIATRIC ENDOCRINOLOGY VZW/ASBL)
Record Dates: First submitted 2016-04-25; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Puberty, Precocious; Adiposity
Keywords: Body Mass Index; Body Composition; Glucose Metabolism Disorders; Bone Development; Gonadal Disorders; Fertility; Overweight; Obesity; Menarche
MeSH Terms: conditions — Puberty, Precocious; Obesity; Glucose Metabolism Disorders; Gonadal Disorders; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GnRHas - Not GnRHas patients (Other): Compared long term outcome of treated and untreated patients with idiopathic central precocious puberty : hormonal assessment; DNA for candidate single nucleotide polymorphisms (SNP) analyses; pelvic ultrasound; dual energy x-ray absorptiometry (DXA)
  Interventions: Other: GnRHas
- GnRHas - controls patients (Other): Compared long term outcome of treated patients with idiopathic central precocious puberty and control patients for: hormonal assessment; DNA for candidate single nucleotide polymorphisms (SNP) analyses; pelvic ultrasound; dual energy x-ray absorptiometry (DXA)
  Interventions: Other: GnRHas
- Not GnRHas - Controls patients (Other): Compared long term outcome of untreated patients with idiopathic central precocious puberty and control patients for: hormonal assessment; DNA for candidate single nucleotide polymorphisms (SNP) analyses; pelvic ultrasound; dual energy x-ray absorptiometry (DXA)
  Interventions: Other: GnRHas

INTERVENTIONS:
Other: GnRHas — Influence of early adiposity rebound, genetic polymorphisms and GnRHa treatment on long-term outcome of treated and untreated girls with idiopathic central precocious compared to a control group.
  puberty.

SUMMARY:
This study evaluates the influence of early adiposity rebound, genetic polymorphisms and GnRHa treatment on long-term outcome of girls with idiopathic central precocious puberty.

DETAILED DESCRIPTION:
Gonadotropin-releasing hormone (GnRH) analogs are the mainstay of treatment for central precocious puberty (CPP) since 1985. The relatively short time period elapsed since the introduction of this therapy has not allowed until now to carry out exhaustive studies on the long-term evolution of treated patients. This project will analyze the long-term outcomes of patients with CPP treated or not with GnRHas on adult height, body mass index, body composition, metabolic disorders, bone mineralization, gonadal function, and fertility in comparison to a control group. Overweight before puberty is associated to earlier menarche, and conversely, earlier menarche predispose to adult obesity and metabolic disorders. Nevertheless, it is unclear if adult adiposity is a direct consequence of early puberty or if early puberty is a marker of a predisposition to excess adiposity from prepuberty through adult life. Recent data in rodent models support the hypothesis that early nutritional status determines a risk for both childhood and adult obesity and influences pubertal timing. In girls, early weight gain in childhood has been associated with early menarche. Pattern of growth rather than absolute level of fatness seem to be of most importance. So the first aim of this study is to compare the outcomes of CCP patients with or without an early adiposity rebound and to demonstrate that adiposity rebound more than CPP per se or the GnRHas therapy affect the outcomes. Moreover, recent genome-wide association studies have identified obesity-related gene variants associated with earlier age at menarche. The investigators hypothesized that there might be a genetic basis underlying the early programming of both childhood and adulthood adiposity and puberty timing. The investigators thus aim to determine if those obesity-related gene variants associated with an early but not precocious menarche could also be found in CPP, especially in girls with an early adiposity rebound and if their presence may affect adult health.

ELIGIBILITY:
Inclusion Criteria:

* History of idiopathic CPP (ICPP) treated with GnRHas.
* A diagnosis of CPP made according to the following criteria: 1) secondary pubertal signs (Tanner stage 2) before 8 years in girls and 9 years in boys; 2) accelerated growth velocity (GV); 3) BA advanced for CA ≥ 1 year; 4) GnRH-stimulated peak LH >5 IU/L.
* A diagnosis of idiopathic CPP according the following criteria: 1) no hypothalamic-pituitary organic lesions at magnetic resonance imaging; 2) no known medical condition that might affect the onset of puberty.
* To determine whether the supposed long-term effects of treatment are instead consequences of the disease itself, untreated ICPP girls aged of ≥ 18 years, will also be included. For comparative purposes, age-matched normal (menarche > 10 y) volunteers will be recruited as a control group.

Exclusion Criteria:

* In the treated ICCP group if 1) treatment with GnRHas for < 2 years; 2) non-compliance; 3) no gonadotropin suppression observed.
* For all patients: 4) small for gestational age; 5) chronic disease and/or treatment; 6) being < 4 years from menarche.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Single nucleotide polymorphisms (SNP) analyses | 1 day
  DNA analyses

SECONDARY OUTCOMES:
Adult height in meters | 1 day
  Measured at consultation
Body mass index in kg/m2 | 1 day
  Calculated at consultation
Body composition in % | 1 day
  Dual energy x-ray absorptiometry (DXA): fat (visceral) and lean mass.
Glucose in mg/dl | 1 day
  Fasting blood sampling
Total Cholesterol in mg/dl | 1 day
  Fasting blood sampling
LDL-Cholesterol in mg/dl | 1 day
  Metabolic assessment (fasting blood sampling)
HDL-Cholesterol in mg/dl | 1 day
  Fasting blood sampling
Insulin in microU/ml | 1 day
  Fasting blood sampling
Total bone mineralization in Tscore | 1 day
  Dual energy x-ray absorptiometry (DXA):
Lumbar bone mineralization in Tscore | 1 day
  Dual energy x-ray absorptiometry (DXA):
Femoral neck bone mineralization in Tscore | 1 day
  Dual energy x-ray absorptiometry (DXA):
Ovaries volume in ml | 1 day
  Pelvic ultrasound (at 2nd-5th day of the menstrual cycle)
Ovaries follicles diameter in mm | 1 day
  Pelvic ultrasound (at 2nd-5th day of the menstrual cycle)
Chronic anovulation in number | 1 day
  Number of mentruals cycles in a year
SHBG by nmol/l | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
Total serum testosterone by ng/dl | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
Ovaries follicles counting | 1 day
  Pelvic ultrasound (at 2nd-5th day of the menstrual cycle)
Abdominal perimeter in cm | 1 day
  Measured at consultation
Hip perimeter in cm | 1 day
  Measured at consultation
Blood pressure in mmHg | 1 day
  Measured at consultation
Testicular volume in ml | 1 day
  Measured at consultation
LH in IU/L | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
FSH in IU/L | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
Oestradiol in ng/dl | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
DHEAS in micromol/l | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
17 hydroxyprogesterone in ng/ml | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
Anti-Müllerian Hormone in ng/ml | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
Inhibine in pg/ml | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
Prolactine in microgr/L | 1 day
  Metabolic assessment (blood sampling before 10 am at the 2nd-5th day of the menstrual cycle or after 2 months of amenorrhea)
Uterine diameter in mm | 1 day
  Pelvic ultrasound (at 2nd-5th day of the menstrual cycle)
Uterine volume in ml | 1 day
  Pelvic ultrasound (at 2nd-5th day of the menstrual cycle)
Endometrius thickness in mm | 1 day
  Pelvic ultrasound (at 2nd-5th day of the menstrual cycle)

OTHER OUTCOMES:
Quality of life | 1 day
  Self-perception profile for adults, Messer & Harter 2012

CONTACTS AND LOCATIONS:
Overall Officials: Constanza Navarro Moreno, D, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for some outcome measures will be made available within 6 months of study recruitment for the Belgian Study Group for Pediatric Endocrinology.

REFERENCES:
- [Background] Lee JM, Appugliese D, Kaciroti N, Corwyn RF, Bradley RH, Lumeng JC. Weight status in young girls and the onset of puberty. Pediatrics. 2007 Mar;119(3):e624-30. doi: 10.1542/peds.2006-2188. PMID 17332182
- [Background] Lakshman R, Forouhi NG, Sharp SJ, Luben R, Bingham SA, Khaw KT, Wareham NJ, Ong KK. Early age at menarche associated with cardiovascular disease and mortality. J Clin Endocrinol Metab. 2009 Dec;94(12):4953-60. doi: 10.1210/jc.2009-1789. Epub 2009 Oct 30. PMID 19880785
- [Background] Parent AS, Franssen D, Fudvoye J, Pinson A, Bourguignon JP. Current Changes in Pubertal Timing: Revised Vision in Relation with Environmental Factors Including Endocrine Disruptors. Endocr Dev. 2016;29:174-84. doi: 10.1159/000438885. Epub 2015 Dec 17. PMID 26680578
- [Background] Sorensen K, Mouritsen A, Aksglaede L, Hagen CP, Mogensen SS, Juul A. Recent secular trends in pubertal timing: implications for evaluation and diagnosis of precocious puberty. Horm Res Paediatr. 2012;77(3):137-45. doi: 10.1159/000336325. Epub 2012 Apr 12. PMID 22508036
- [Background] Copeland W, Shanahan L, Miller S, Costello EJ, Angold A, Maughan B. Outcomes of early pubertal timing in young women: a prospective population-based study. Am J Psychiatry. 2010 Oct;167(10):1218-25. doi: 10.1176/appi.ajp.2010.09081190. Epub 2010 May 17. PMID 20478880
- [Background] Carel JC, Eugster EA, Rogol A, Ghizzoni L, Palmert MR; ESPE-LWPES GnRH Analogs Consensus Conference Group; Antoniazzi F, Berenbaum S, Bourguignon JP, Chrousos GP, Coste J, Deal S, de Vries L, Foster C, Heger S, Holland J, Jahnukainen K, Juul A, Kaplowitz P, Lahlou N, Lee MM, Lee P, Merke DP, Neely EK, Oostdijk W, Phillip M, Rosenfield RL, Shulman D, Styne D, Tauber M, Wit JM. Consensus statement on the use of gonadotropin-releasing hormone analogs in children. Pediatrics. 2009 Apr;123(4):e752-62. doi: 10.1542/peds.2008-1783. Epub 2009 Mar 30. PMID 19332438
- [Background] Klein KO, Barnes KM, Jones JV, Feuillan PP, Cutler GB Jr. Increased final height in precocious puberty after long-term treatment with LHRH agonists: the National Institutes of Health experience. J Clin Endocrinol Metab. 2001 Oct;86(10):4711-6. doi: 10.1210/jcem.86.10.7915. PMID 11600530
- [Background] Brito VN, Latronico AC, Cukier P, Teles MG, Silveira LF, Arnhold IJ, Mendonca BB. Factors determining normal adult height in girls with gonadotropin-dependent precocious puberty treated with depot gonadotropin-releasing hormone analogs. J Clin Endocrinol Metab. 2008 Jul;93(7):2662-9. doi: 10.1210/jc.2007-2183. Epub 2008 May 6. PMID 18460564
- [Background] Lazar L, Lebenthal Y, Yackobovitch-Gavan M, Shalitin S, de Vries L, Phillip M, Meyerovitch J. Treated and untreated women with idiopathic precocious puberty: BMI evolution, metabolic outcome, and general health between third and fifth decades. J Clin Endocrinol Metab. 2015 Apr;100(4):1445-51. doi: 10.1210/jc.2014-3748. Epub 2015 Feb 4. PMID 25650898
- [Background] Magiakou MA, Manousaki D, Papadaki M, Hadjidakis D, Levidou G, Vakaki M, Papaefstathiou A, Lalioti N, Kanaka-Gantenbein C, Piaditis G, Chrousos GP, Dacou-Voutetakis C. The efficacy and safety of gonadotropin-releasing hormone analog treatment in childhood and adolescence: a single center, long-term follow-up study. J Clin Endocrinol Metab. 2010 Jan;95(1):109-17. doi: 10.1210/jc.2009-0793. Epub 2009 Nov 6. PMID 19897682
- [Background] Franceschi R, Gaudino R, Marcolongo A, Gallo MC, Rossi L, Antoniazzi F, Tato L. Prevalence of polycystic ovary syndrome in young women who had idiopathic central precocious puberty. Fertil Steril. 2010 Mar 1;93(4):1185-91. doi: 10.1016/j.fertnstert.2008.11.016. Epub 2009 Jan 9. PMID 19135667
- [Background] Barker DJ, Osmond C, Forsen TJ, Kajantie E, Eriksson JG. Trajectories of growth among children who have coronary events as adults. N Engl J Med. 2005 Oct 27;353(17):1802-9. doi: 10.1056/NEJMoa044160. PMID 16251536
- [Background] Brockenbrough JS, Meyer SA, Li CX, Jirtle RL. Reversible and phorbol ester-specific defect of protein kinase C translocation in hepatocytes isolated from phenobarbital-treated rats. Cancer Res. 1991 Jan 1;51(1):130-6. PMID 1988078
- [Background] Canoy D, Beral V, Balkwill A, Wright FL, Kroll ME, Reeves GK, Green J, Cairns BJ; Million Women Study Collaborators*. Age at menarche and risks of coronary heart and other vascular diseases in a large UK cohort. Circulation. 2015 Jan 20;131(3):237-44. doi: 10.1161/CIRCULATIONAHA.114.010070. Epub 2014 Dec 15. PMID 25512444
- [Background] Colmenares A, Gunczler P, Lanes R. Higher prevalence of obesity and overweight without an adverse metabolic profile in girls with central precocious puberty compared to girls with early puberty, regardless of GnRH analogue treatment. Int J Pediatr Endocrinol. 2014;2014(1):5. doi: 10.1186/1687-9856-2014-5. Epub 2014 Apr 17. PMID 24742263
- [Background] Ibanez L, Lopez-Bermejo A, Diaz M, Suarez L, de Zegher F. Low-birth weight children develop lower sex hormone binding globulin and higher dehydroepiandrosterone sulfate levels and aggravate their visceral adiposity and hypoadiponectinemia between six and eight years of age. J Clin Endocrinol Metab. 2009 Oct;94(10):3696-9. doi: 10.1210/jc.2009-0789. Epub 2009 Sep 8. PMID 19737922
- [Background] Dreyfus J, Jacobs DR Jr, Mueller N, Schreiner PJ, Moran A, Carnethon MR, Demerath EW. Age at Menarche and Cardiometabolic Risk in Adulthood: The Coronary Artery Risk Development in Young Adults Study. J Pediatr. 2015 Aug;167(2):344-52.e1. doi: 10.1016/j.jpeds.2015.04.032. Epub 2015 May 9. PMID 25962931
- [Background] Clark EM, Ness AR, Tobias JH. Adipose tissue stimulates bone growth in prepubertal children. J Clin Endocrinol Metab. 2006 Jul;91(7):2534-41. doi: 10.1210/jc.2006-0332. Epub 2006 Apr 18. PMID 16621904
- [Background] Yanovski JA, Rose SR, Municchi G, Pescovitz OH, Hill SC, Cassorla FG, Cutler GB Jr. Treatment with a luteinizing hormone-releasing hormone agonist in adolescents with short stature. N Engl J Med. 2003 Mar 6;348(10):908-17. doi: 10.1056/NEJMoa013555. PMID 12621135
- [Background] Chiavaroli V, Liberati M, D'Antonio F, Masuccio F, Capanna R, Verrotti A, Chiarelli F, Mohn A. GNRH analog therapy in girls with early puberty is associated with the achievement of predicted final height but also with increased risk of polycystic ovary syndrome. Eur J Endocrinol. 2010 Jul;163(1):55-62. doi: 10.1530/EJE-09-1102. Epub 2010 Mar 31. PMID 20356934
- [Background] Ong KK, Elks CE, Wills AK, Wong A, Wareham NJ, Loos RJ, Kuh D, Hardy R. Associations between the pubertal timing-related variant in LIN28B and BMI vary across the life course. J Clin Endocrinol Metab. 2011 Jan;96(1):E125-9. doi: 10.1210/jc.2010-0941. Epub 2010 Oct 20. PMID 20962026
- [Background] Conway G, Dewailly D, Diamanti-Kandarakis E, Escobar-Morreale HF, Franks S, Gambineri A, Kelestimur F, Macut D, Micic D, Pasquali R, Pfeifer M, Pignatelli D, Pugeat M, Yildiz BO; ESE PCOS Special Interest Group. The polycystic ovary syndrome: a position statement from the European Society of Endocrinology. Eur J Endocrinol. 2014 Oct;171(4):P1-29. doi: 10.1530/EJE-14-0253. Epub 2014 May 21. PMID 24849517
- [Background] Deb S, Campbell BK, Pincott-Allen C, Clewes JS, Cumberpatch G, Raine-Fenning NJ. Quantifying effect of combined oral contraceptive pill on functional ovarian reserve as measured by serum anti-Mullerian hormone and small antral follicle count using three-dimensional ultrasound. Ultrasound Obstet Gynecol. 2012 May;39(5):574-80. doi: 10.1002/uog.10114. PMID 21997961